CLINICAL TRIAL: NCT04775680
Title: A Multicenter, Open-Label, Phase Ib/II Study of ADG106 in Combination With PD-1 Antibody in Advanced Solid Tumors and Relapsed/Refractory Non-Hodgkin Lymphoma
Brief Title: Study of ADG106 In Combination With PD-1 Antibody In Advanced or Metastatic Solid Tumors and/or Non Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The safety of ADG106 combined with triprilimab has been fully understood.The overall clinical benefit of enrolled subjects was limited and further development of ADG106 was reconsidered.
Sponsor: Adagene (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Organization: Adagene Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADG106-1008
Record Dates: First submitted 2021-02-16; First posted 2021-03-01 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Solid Tumor; Non Hodgkin Lymphoma
Keywords: Solid Tumor and Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADG106 combined with PD-1 antibody Dose Escalation Level 1 (Experimental)
  Interventions: Biological: ADG106 injection; Biological: PD-1 antibody injection
- ADG106 combined with anti PD-1 antibody Dose Escalation Level 2 (Experimental)
  Interventions: Biological: ADG106 injection; Biological: PD-1 antibody injection
- ADG106 combined with anti PD-1 antibody Expansion Phase (Experimental)
  Interventions: Biological: ADG106 injection; Biological: PD-1 antibody injection

INTERVENTIONS:
Biological: ADG106 injection — ADG106 injection, intravenous infusion, is administered as body weight every 3 weeks for 21 days as a cycle
Biological: PD-1 antibody injection — PD-1 antibody injection is administered as an intravenous infusion and at a dose of 240mg every 3 weeks for 21 days as a cycle

SUMMARY:
This is a Multicenter, Open-Label, Phase Ib/II Study of ADG106 in Combination with PD-1 Antibody in Advanced Solid Tumors and Relapsed/Refractory Non-Hodgkin Lymphoma.

The primary objective of Phase Ib: To evaluate the maximum tolerated dosage (MTD) of ADG106 in combination with PD-1 antibody in advanced solid tumors and relapsed/refractory non-Hodgkin lymphoma, and to determine the recommended phase II clinical studies dosage (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced solid tumors or relapses/refractory non-Hodgkin's lymphoma confirmed by histology or cytology
* Has at least one measurable lesion (solid tumor according to RECIST v1.1 criteria, non-Hodgkin's lymphoma according to Lugnao criteria)
* ECOG score of 0 or 1;
* Expected survival time ≥ 3 months (at the discretion of the investigator);
* Adequate organ and bone marrow function;
* Voluntarily sign the informed consent form;

Exclusion Criteria:

* Has central nervous system primary malignant tumor, active epileptic seizure, spinal cord compression or carcinomatous meningitis
* The previous anti-tumor treatment has not passed the prescribed washout period
* HIV antibody is positive, or with other acquired/congenital immunodeficiency disease, or with history of organ transplantation;
* Active hepatitis B or hepatitis C virus (HCV) antibody was positive;
* Patients who are pregnant or lactating;
* Known or suspected hypersensitivity to the study drug or its pharmaceutical excipients (including mono-hydrate citric acid, sodium di-hydrate citric acid, mannitol, polysorbate, arginine, succinic acid);
* Any active autoimmune disease, or known history of autoimmune disease, or syndrome requiring systemic steroids or immunosuppressive medications (other than controlled thyroid disease with alternative therapy/non-immunosuppressive therapy);
* Participation in another therapeutic or interventional clinical study in the meantime;
* Other circumstances where the investigator considers it is not appropriate to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing dosage limiting toxicity (DLT) in the first treatment cycle of the combination of ADG106 and PD-1 antibody. | From first dose of ADG106 and PD-1 antibody (Week 1 Day 1) until 21 days
Objective response rate (ORR) of the combination of ADG106 and PD-1 antibody in advanced solid tumors and relapsed/refractory non-hodgkin lymphoma | From baseline to measured progressive disease (up to 24 months)

SECONDARY OUTCOMES:
Type of adverse event, incidence, grade (according to NCI CTCAE V 5.0 classification), onset time, and relationship to study treatment | From the first dose of ADG106 and PD-1 antibody (Week 1 Day 1) to 28 days post last dose
Area under the time concentration curve(AUC) from time zero to infinity (AUC0-inf)) | From the first dose of ADG106 and PD-1 antibody (Cycle 1 Day 1,each cycle is 21 days) until the last dose (up to 2 years)
Maximum (peak) plasma concentration (Cmax) | From the first dose of ADG106 and PD-1 antibody (Cycle 1 Day 1,each cycle is 21 days) until the last dose (up to 2 years)
Time to maximum(peak) plasma concentration Tmax | From the first dose of ADG106 and PD-1 antibody (Cycle 1 Day 1,each cycle is 21 days) until the last dose (up to 2 years)
Through plasma concentration(Cthrough) | From the first dose of ADG106 and PD-1 antibody (Cycle 1 Day 1,each cycle is 21 days) until the last dose (up to 2 years)
Anti-drug antibody levels of ADG106 and PD-1 antibody | From the first dose of ADG106 and PD-1 antibody (Cycle 1 Day 1,each cycle is 21 days) until the last dose (up to 2 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No